CLINICAL TRIAL: NCT06858163
Title: Coping and Attachment in Pediatric Oncohematology: Multicenter Cross-sectional Study to Assess Emotional Resources and Attachment Dynamics Related to Coping Strategies in Parents of Children with Oncohematologic Disease
Brief Title: Coping and Attachment in Pediatric Oncohematology
Acronym: CopAt
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Fondazione Soleterre - Strategie di Pace ONLUS (Unknown); Università Pavia - Dipartimento di Scienze del Sistema Nervoso e del Comportamento (Unknown); Università Cattolica Milano - Unità di ricerca sul Trauma, Dipartimento di Psicologia (Unknown)
Responsible Party: Principal Investigator, Marco Zecca, Head of Pediatric Oncohematology department, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: CopAt
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Cancer; Coping Behavior; Relationship, Parent Child
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Parents cohort: Father and mother of each patient in care at the Pediatric Oncohematology department and enrolled in the study.
  The correlation between attachment dynamics and emotional care resources related to coping strategies will be assessed.
  Administration of psychological tests will take place one time after the enrollment in the study.
- Patients cohort: Pediatric patients in care at the Pediatric Oncohematology department. Administration of psychological tests will take place one time after the enrollment in the study.

SUMMARY:
Cancer can be a traumatic and particularly salient experience in a person's history. The ways in which the pediatric patient copes with it depend on the interaction of several factors present in his or her life context, primarily the relationship that is established between parent and child.

Despite the paucity of studies in the literature in this regard, it would seem that parental coping is predictive of child coping. Coping strategies represent the ways in which people try to manage traumatic events or stressful everyday situations.

Currently, the literature identifies two main categories of coping strategies: emotion-oriented and problem-oriented strategies. The former are aimed on reducing stress-induced unpleasant emotions (e.g., problem avoidance, positive reappraisal, etc.); the latter, on the other hand, focus on stress dissolution/alteration (e.g., problem identification and resolution, stress cause research). Some studies, previously conducted in oncology, show that emotion-focused coping strategies are associated with better adaptation immediately after diagnosis, but their positive influence tends to weaken over time; problem-focused coping strategies are more correlated with poor adaptation immediately after diagnosis, but in the later stages of treatment.

The clinical experience with patients in the Pediatric Oncohematology Department brings out the need to develop and structure a psychological assessment model, in order to ensure a more effective care of the family units followed.

The research aims, through a single administration of psychological tests, to investigate the role of attachment and some variables (age, gender, stage of treatment, stage of the disease, social support, resilience, ability to adapt to environmental stimuli, emotional state of of caregivers) on the coping strategies implemented by the parents of patients and the patients themselves, in order to differentiate the types of psychological intervention, to try to reduce psychological distress and increase levels of mental well-being.

ELIGIBILITY:
Parents Inclusion Criteria:

* parents of both sexes
* age of son/daughter between 8 and 17 years old (included)
* son/daughter being treated at the Pediatric Oncohematology departments involved in the research (Day Hospital and hospitalization)
* good understanding of the Italian language

Parents Exclusion Criteria:

● son/daughter in off-therapy

Patients Inclusion Criteria:

* age between 8 and 17 years old (included), undergoing treatment at the Pediatric Oncohematology departments (Day Hospital and hospitalization)
* parents enrolled in the study
* good understanding of the Italian language

Patients Exclusion Criteria:

● patients in off-therapy

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Parents (single/father and mother) of patients in care of Pediatric Oncohematology departments who meet the inclusion criteria and pediatric patients in treatment at the Pediatric Oncohematology departments who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Child-Parent Relationship Scale | One time just after the enrollment
  Child-Parent Relationship Scale is a 30-item, self-report instrument used to assess conflict and relational closeness, two important aspects in the emotional support provided to the child and compliance with care, as well as perceived parental distress. The Likert scale ranges from 1 to 5, where 1 stands for "Absolutely not true" and 5 stands for "Definitely true." Scoring is done by summing the raw scores of the items in the three sections (positive aspects of the relationship, conflict and dependence) divided by the items in each sub-scale (mean score).
Coping Orientations to Problem Experienced | One time just after the enrollment
  "Coping Orientations to Problem Experienced- New Italian Version" is a self-report questionnaire that considers different coping modes. The Likert scale ranges from 1 to 4, where 1 stands for "I usually don't do it" and 4 stands for "I almost always do it." The instrument consists of 60 items, divided into 5 independent dimensions: social support, avoidance strategies, positive attitude, problem orientation and transcendent orientation. The scores from 1 to 4 are based on the responses identified by the subject for each item except for 4 "reverse" responses (items 8-20-36-50) for which the chosen score must be reversed. The items are then divided into groups for the identification of the 5 coping factors (social support, avoidance, positive attitude and transcendent orientation). Higher scores indicate greater use of that specific coping strategy.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Ospedale San Gerardo, SC Ematologia Pediatrica, Monza, Monza-Brianza
  - SC Ematologia 2 - Oncoematologia pediatrica, Pavia, Pavia
  - Struttura Complessa di Pediatria e Oncoematologia Pediatrica, Ospedale SS Annunziata, Taranto, Taranto

REFERENCES:
- [Background] Lazarus, R. S., and Folkman, S. (1984). Stress, Appraisal and Coping. New York, NY: Springer.
- [Background] Sica, C., Magni, C., Ghisi, M., Altoè, G., Sighinolfi, C., Chiri, L. R., & Franceschini, S. (2008). Coping Orientation to Problems Experienced-Nuova Versione Italiana (COPE-NVI): uno strumento per la misura degli stili di coping. Psicoterapia cognitiva e comportamentale, 14(1), 27.
- [Background] Monti JD, Winning A, Watson KH, Williams EK, Gerhardt CA, Compas BE, Vannatta K. Maternal and Paternal Influences on Children's Coping with Cancer-Related Stress. J Child Fam Stud. 2017 Jul;26(7):2016-2025. doi: 10.1007/s10826-017-0711-y. Epub 2017 Apr 17. PMID 29056838